CLINICAL TRIAL: NCT01797471
Title: A Phase 1 Study for Evaluating the Safety of Lattice Extreme Ablative Dose (LEAD) Radiotherapy Followed by Standard-Dose Chemoradiation for Patients With Bulky Stage III Non-Small Cell Lung Cancer
Brief Title: Safety of LEAD Radiotherapy Plus Chemoradiation in Patients With Bulky Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100446
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Non-Small Cell Lung Cancer; NSCLC
Keywords: Non-Small Cell Lung Cancer; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Lead; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LEAD RT (Experimental): * Lattice Extreme Ablative Dose (LEAD) Radiation Therapy (RT) on Day 1 at dose of 18 Gy followed by;
  * Conventionally fractionated radiation therapy beginning on day 2 at 2 Gy per fraction for 30 fractions for a total dose of 60 Gy;
  * Conventional Platinum Chemotherapy Doublet at discretion of treating physician beginning on day 2.
  Interventions: Radiation: Lattice Extreme Ablative Dose (LEAD) Radiation Therapy

INTERVENTIONS:
Radiation: Lattice Extreme Ablative Dose (LEAD) Radiation Therapy — A single fraction of LEAD RT, dose of 18 Gy will be delivered to subjects on day 1
  Other Names: LEAD Radiotherapy; LEAD Radiation Therapy

SUMMARY:
The investigators aim to evaluate the safety of delivering a one-time single fraction of Lattice Extreme Ablative Dose (LEAD) radiotherapy followed one day later by standard-dose, conventionally fractionated concurrent chemotherapy and radiation delivered over 6 weeks in patients with bulky stage III non-small cell lung cancer in the setting of a single-arm phase I clinical trial. The investigators hypothesize that the addition of a one-time single fraction of LEAD radiation is safe and feasible, and will not result in additional toxicity above that expected with standard-dose concurrent chemotherapy and radiation alone.

DETAILED DESCRIPTION:
Paarticipants will receive a single fraction of LEAD radiation on day 1, followed one day later by conventionally fractionated concurrent chemoradiation consisting of 60 Gy of radiation delivered to involved sites of disease and a platinum doublet.

The investigational radiation treatment, a single fraction of LEAD radiation, is to be followed by conventionally fractionated radiation delivered concurrently with a standard chemotherapy regimen for stage III non-small cell lung cancer. The following day, patients will begin concurrent chemotherapy and radiation. Chemotherapy will be delivered under the management of the treating medical oncologist. Chemotherapy must be a platinum doublet. Carboplatin and cisplatin are both considered acceptable platinum agents. The use of cisplatin over carboplatin is strongly encouraged, unless the patient has a contraindication to cisplatin. The second agent will be at the discretion of the treating medical oncologist; in the current era, chemotherapy agents are tailored to each patient based on tumor histology, as well as comorbidities that dictate the tolerance of certain chemotherapeutic agents. Chemotherapy will be delivered concurrently throughout radiation therapy, beginning on day 2 of the treatment protocol and on the same day as the start of standard-dose radiation. Weekly regimens or regimens delivered every 3 weeks are acceptable. Additional cycles of consolidation chemotherapy are encouraged and will be given at the discretion of the treating medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically documented stage III non-small cell lung cancer including squamous cell, adenocarcinoma, large cell carcinoma and poorly differentiated non-small cell lung cancer.
2. Patients must have a minimum of 4 cm of measurable disease in any one continuous dimension as seen on diagnostic CT scan.
3. Pulmonary function tests with forced expiratory volume in 1 second (FEV1) ≥1.45 liters/second.
4. Patients must be 21 years of age or older. There is no maximum age restriction.
5. Patients must have a Zubrod performance status of 0 or 1.
6. Patients must have normal organ and marrow function as defined below:

   * leukocyte > 3,000/:I
   * absolute neutrophil count >1,500/:I
   * platelets >100,000/:I
   * bilirubin within normal institutional limits
   * Aspartate transaminase (AST/SGOT)/Alanine transaminase (ALT/SGPT) 2.5 X institutional upper limit of normal
   * Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
7. Patients must have weight loss ≤ 10% over the past three months.
8. Women of child-bearing potential and men will be asked to use adequate contraception.
9. Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients may not have had prior thoracic radiation at any time, or prior chemotherapy for the study cancer at any time.
2. Patients may not be receiving any other investigational agents for the study cancer.
3. Patients may not have evidence of brain metastases on baseline CT scan or MRI.
4. Patients may not have measurable gross disease in the thorax <4 cm in any one continuous dimension.
5. Patients may not have a cytologically positive pleural effusion.
6. Patients may not have a prior invasive malignancy (unless disease-free for at least 3 years).
7. Patients may not have had surgical resection of the present cancer.
8. Women who are pregnant or breastfeeding will be excluded.
9. Patients must not have any co-morbidity with life expectancy ≤ 6 months, or any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patients must not have severe lung disease defined by a history of severe chronic obstructive pulmonary disease (COPD) requiring 3 or more hospitalizations over the past year, or history of interstitial pneumonitis.
11. Patients must not have any concurrent active malignancy.
12. Patients must not have evidence of metastatic disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05-31 (Actual); Study Completion 2013-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Wright, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LEAD RT: * Lattice Extreme Ablative Dose Radiation Therapy (RT) on Day 1 at dose of 18 Gy followed by;
  * Conventionally fractionated radiation therapy beginning on day 2 at 2 Gy per fraction for 30 fractions for a total dose of 60 Gy;
  * Conventional Platinum Chemotherapy Doublet at discretion of treating physician beginning on day 2.
  Lattice Extreme Ablative Dose Radiation Therapy: A single fraction of LEAD RT, dose of 18 Gy will be delivered to subjects on day 1
Period: Overall Study
Arm/Group | LEAD RT
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LEAD RT
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Treatment-related Toxicity in Study Participants
Description: Rate of treatment-related toxicity (serious adverse events, adverse events, etc.) in study participants. Toxicity will be assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The two toxicities that will be monitored as primary endpoints are esophagitis and pneumonitis.
Time Frame: Up to 12 months
Population: Study participants experiencing treatment-related esophagitis or pneumonitis.
Measure: Count of Participants; unit: Participants
Arm/Group | LEAD RT
Number analyzed (Participants) | 1
Participants
  Esophagitis | 1
  Pneumonitis | 0

2. Secondary Outcome: Rate of Study Participants Achieving Complete or Partial Response Via CT RECIST Response Criteria
Description: Number of subjects achieving complete response (CR) or partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria on CT Scan:
  * CR: Complete disappearance of all disease. No new lesions. No disease related symptoms. Normalization of markers and other abnormal lab values. All disease must be assessed using the same technique as baseline.
  * PR: Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions.
Time Frame: Assessed up to 2 years
Population: A minimum sample size of 10 study participants was required for the analysis of the outcome. Minimum enrollment was not met, therefore, the data were not analyzed.
Arm/Group | LEAD RT
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Study Participants Achieving Complete or Partial Response Via PET Response Criteria
Description: Rate of subjects achieving complete response (CR) or partial response (PR) as detected by positron emission tomography (PET) Scan:
  * CR is defined as no residual focal fluorodeoxyglucose (FDG) uptake or decrease in average FDG uptake by more than 80% in all tumor manifestations.
  * PR is defined as standardized uptake value (SUV) decrease by 0 - 80%.
Time Frame: Assessed up to 2 years
Population: A minimum sample size of 10 study participants was required for the analysis of the outcome measure. Minimum enrollment was not met, therefore, the data were not analyzed.
Arm/Group | LEAD RT
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Loco-regional Failure in Study Participants
Description: Rate of loco-regional failure in study participants. Loco-regional failure is defined as any evidence of disease progression within the primary primary tumor or regional lymph nodes, detected by any method.
Time Frame: Assessed up to 2 years
Population: as for outcome 3
Arm/Group | LEAD RT
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Rate of progression-free survival (PFS). PFS is defined as the length of time from date of treatment initiation until date of documented disease progression or death from any cause, with censoring of patients who are lost to follow-up.
Time Frame: Assessed up to 2 years
Population: as for outcome 3
Arm/Group | LEAD RT
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Rate of overall survival (OS) in study participants. Overall survival is defined as the length of time from the date of treatment initiation until the date of death from any cause.
Time Frame: Assessed up to 2 years
Population: as for outcome 3
Arm/Group | LEAD RT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | LEAD RT
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEAD RT (N=1)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEAD RT (N=1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A minimum sample size of 10 study participants was required for the analysis of most outcome measures. Minimum enrollment was not met, therefore, the data for these applicable outcome measures were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes